CLINICAL TRIAL: NCT05276908
Title: Analgesic Efficacy of Two Different Volumes of Local Anesthetics in Ultrasound-guided Modified Approach of Thoracolumbar Block in Patients Undergoing Lumbar Spine Surgeries; a Randomized Controlled Trial.
Brief Title: Different Volumes of Local Anesthetics in Thoracolumbar Interfascial Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, Assissnt professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-307-2020
Record Dates: First submitted 2022-02-28; First posted 2022-03-14 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mTLIP10 (Experimental): patients will receive single shot of bilateral modified thoracolumbar interfascial plane block at the mid-level of the operative intervention with 20 ml 0.25%bupivacaine (10 ml on each side).
  Interventions: Procedure: Thoracolumbar interfascial plane block (TLIP)Technique; Procedure: Anesthetic Management; Drug: Bupivacaine Injection 10ml
- mTLIP20 (Experimental): patients will receive single shot of bilateral modified thoracolumbar interfascial plane block at the mid-level of the operative intervention with 40 ml 0.25%bupivacaine (20 ml on each side).
  Interventions: Procedure: Thoracolumbar interfascial plane block (TLIP)Technique; Procedure: Anesthetic Management; Drug: Bupivacaine Injection 20ml

INTERVENTIONS:
Procedure: Thoracolumbar interfascial plane block (TLIP)Technique — A curvilinear array ultrasound probe (Siemens ACUSON X300 Ultrasound System) will be placed at the targeted lumbar level.The corresponding spinous process and interspinal muscles will be identified, and the probe will be slided laterally to identify the longissimus muscle and iliocostalis muscle. Under ultrasound guidance, A 38-mm 22-gauge (22-G, 50-mm 'Stimuplex; BBraun, Melsung, Germany) regional block needle will be advanced in plane to the ultrasound beam in a medial to lateral orientation through the belly of longissimus muscle toward the iliocostalis muscle. Hydro-dissection with 2-3 ml of isotonic saline solution will confirm the correct needle tip position and, after negative aspiration, 0.25 % bupivacaine will be injected slowly whilst carefully monitoring the spread of local anesthetic into the fascial plane between the longissimus and iliocostalis muscles. The same procedure will be repeated on the contralateral side.
Procedure: Anesthetic Management — Induction:
  Induction of general anesthesia will be performed using a regimen of IV 2 μg/kg fentanyl and propofol IV 2 mg /kg. Tracheal intubation will be facilitated using 0.5 mg/kg IV of atracurium.
  Maintenance:
  Anesthesia will be maintained with inhaled isoflurane 0.8% in oxygen enriched air (FiO2=0.5). Maintenance doses of 0.1 m\kg atracurium will be provided every 30 minutes. Then the patient will be placed in prone position.
Drug: Bupivacaine Injection 10ml — patients will receive single shot of bilateral modified thoracolumbar interfascial plane block at the mid-level of the operative intervention with 20 ml 0.25%bupivacaine (10 ml on each side).
  Arms: mTLIP10
Drug: Bupivacaine Injection 20ml — patients will receive single shot of bilateral modified thoracolumbar interfascial plane block at the mid-level of the operative intervention with 40 ml 0.25%bupivacaine (20 ml on each side).
  Arms: mTLIP20

SUMMARY:
Ultrasound-guided thoracolumbar interfascial plane block (TLIP)was first described in 2015 by Hand et al which also target the dorsal rami of the thoracolumbar nerves as they pass through the paraspinal musculature(between the multifidus muscle (MF) and the longissimus muscle (LG)). The block was performed bilaterally at the level of L3 and they reported a reproducible area of anesthesia to pinprick in a mean (SD) area covering 137.4 (71.0) cm2 of the lower back (including the midline) after 20 minutes of the block. This procedure has subsequently been modified by Ueshima H et al in 2016 by targeting the injection in the plane between the longissimus and iliocostalis muscles (mTLIP) which helps avoiding the spread of local anesthetics to the ventral ramus and neuraxial space, thus, the modified TLIP block is considered to be a more refined version of the original TLIP block and safer and easier to perform.

There are limited number of studies investigating the analgesic efficacy of mTLIP block however, no previous study has demonstrated the ideal local anesthetic volume for this block in lumber spine surgery. Moreover, this technique is considered new regional anesthetic techniques and so both of them should be involved in further studies, on the other hand the comparison between both of them at the same study wasn't discussed before, and so we will proceed at this study.

DETAILED DESCRIPTION:
The aim of this study is to compare the post-operative analgesic efficacy of two different volumes of local anesthetics in bilateral modified thoracolumbar interfascial plane block in lumbar spine surgeries.

Prospective randomized double blinded study The study will be conducted in Kasr Alainy hospital orthopedic surgical theater. Adult patients undergoing lumbar spine surgeries involving 1 up to 3 adjacent lumbar vertebrae (eg. laminectomy, discectomy …). at Kasr Alainy hospital.

ELIGIBILITY:
Inclusion Criteria:

* ● Both gender

  * Type of surgery: lumbar spine surgeries involving 1 up to 3 adjacent lumbar vertebrae
  * Physical status ASA I, II.
  * Age 18 to 65 Years.
  * Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* ● Patients on preoperative opioid regimen for more than 1 month.

  * Patients with history of previous surgical operations in the lumbar region.
  * Patients with spinal deformities (eg. Scoliosis…..).
  * Hypersensitivity to Bupivacaine.
  * Extensive Lumbar spine surgeries like large tumor excisions, scoliosis correction or more than 2 level spine fixations.
  * Patients with communication difficulties.
  * Lumbar spine operations that will be performed with the patient in any position other than the prone position.
  * Severe neurological compromise (severe muscle weakness such as foot drop or sphincter disorders such as urinary incontinence).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption in the first 24 hours postoperative | 24 hours

SECONDARY OUTCOMES:
Time to first rescue analgesia | 24 hours
  measured from time of block administration to time of rescue analgesia administration
Numeric Pain Rating Scale | 24 hours
  Pain scale of managmet when zero indicates no pain and ten indicates maximum pain both at rest and during movement: 30 minutes,2, 4,6, 8, 12, 16, 20 and 24postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Bassant Abdelhamid, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ammar MA, Taeimah M. Evaluation of thoracolumbar interfascial plane block for postoperative analgesia after herniated lumbar disc surgery: A randomized clinical trial. Saudi J Anaesth. 2018 Oct-Dec;12(4):559-564. doi: 10.4103/sja.SJA_177_18. PMID 30429737
- [Background] Li C, Jia J, Qin Z, Tang Z. The use of ultrasound-guided modified thoracolumbar interfascial plane (TLIP) block for multi-level lumbar spinal surgery. J Clin Anesth. 2018 May;46:49-51. doi: 10.1016/j.jclinane.2018.01.018. Epub 2018 Mar 26. No abstract available. PMID 29414616
- [Derived] Abdelhamid B, Ayman E, Nabil T, Hamimy WI, El-Monem Morsy MA. Analgesic efficacy of two different volumes of local anaesthetics in ultrasound-guided modified approach to the thoracolumbar interfascial plane block in patients undergoing lumbar spine surgeries: a randomized controlled trial. Anaesthesiol Intensive Ther. 2023;55(5):358-365. doi: 10.5114/ait.2023.134196. PMID 38282503